CLINICAL TRIAL: NCT00673374
Title: Correlation of Location of Abdominal Tenderness With Acute CT Abnormalities in Emergency Department Patients
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Principal Investigator, Joshua Broder, Associate Professor, Duke University
Other Study IDs: Pro00004904
Record Dates: First submitted 2008-03-09; First posted 2008-05-07 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Abdominal Pain
Keywords: emergency; acute; nontraumatic; abdominal pain; tenderness; CT scan; radiation; diagnosis
MeSH Terms: conditions — Abdominal Pain; Emergencies; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All consecutive emergency department patients undergoing abdominal CT for non-traumatic abdominal pain and tenderness will be prospectively enrolled, except for those meeting pre-specified exclusion criteria.
  Interventions: Device: radio-opaque adhesive skin markers

INTERVENTIONS:
Device: radio-opaque adhesive skin markers — The examining physician will place a radio-opaque skin marker (Beekley Corporation, Ortho-SPOTS® Order Code 187; 6mm spherical markers) at the point of maximal tenderness to direct abdominal palpation indicated by the patient. Additional markers will be placed at the cephalad and caudad limits of the region of tenderness, defined as the point at which the patient no longer complains of direct tenderness to palpation.

SUMMARY:
To determine the correlation between the region of abdominal tenderness determined by the examining physician and the location of acute pathology diagnosed on abdominal CT. We hypothesize that the acute pathology diagnosed by CT will lie within the region marked on the abdominal wall by the examining physician prior to CT.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive emergency department patients undergoing abdominal CT for non-traumatic abdominal pain and tenderness will be prospectively enrolled, with the following exceptions. For study purposes, "abdominal pain and tenderness" is defined as pain and tenderness to direct palpation in the region anterior to the mid-axillary line bilaterally, and extending from the costal margins to the inguinal ligaments. Consequently, patients undergoing CT for indications such as isolated vomiting, fever without source, staging of malignancies, isolated flank pain or suspected renal colic, or other indications that do not meet the above definition will not be enrolled.

Exclusion Criteria:

* Pregnant women do not routinely undergo abdominal CT due to radiation concerns and will be excluded from the study.
* Patients with altered mental status or altered abdominal sensation (due to neurological conditions such as paraplegia) that may prevent assessment of the location of abdominal tenderness will be excluded.
* Preverbal children will be excluded as they rarely undergo CT and will be unable to indicate the region of maximal tenderness.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive emergency department patients undergoing abdominal CT for non-traumatic abdominal pain and tenderness will be prospectively enrolled, with the following exceptions. For study purposes, "abdominal pain and tenderness" is defined as pain and tenderness to direct palpation in the region anterior to the mid-axillary line bilaterally, and extending from the costal margins to the inguinal ligaments. Consequently, patients undergoing CT for indications such as isolated vomiting, fever without source, staging of malignancies, isolated flank pain or suspected renal colic, or other indications that do not meet the above definition will not be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
sensitivity and specificity of a hypothetical limited CT restricted to the region of abdominal tenderness for detection of acute pathology on CT on the entire abdomen. | immediate

SECONDARY OUTCOMES:
the percentage decrease in radiation exposure which could be achieved by performing a CT restricted to the region of abdominal tenderness, compared with CT of the entire abdomen | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Joshua S Broder, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States